CLINICAL TRIAL: NCT03344250
Title: A Phase I Study Targeting Newly Diagnosed Glioblastoma With Anti-CD3 × Anti-EGFR Bispecific Antibody Armed T Cells (EGFR BATs) in Combination With Radiation and Temozolomide
Brief Title: Phase I EGFR BATs in Newly Diagnosed Glioblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Camilo E. Fadul, MD, Professor, University of Virginia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20105
Record Dates: First submitted 2017-11-02; First posted 2017-11-17 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2023-01

CONDITIONS: Glioblastoma; Glioblastoma Multiforme
Keywords: Adoptive Cell Therapy; Armed Activated T-cells; Bispecific Antibodies; Immunotherapy
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Intervention Model Description: EGFR BATs administered in combination with standard of care temozolomide and radiation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Main Study (Experimental): Study participants will have cells collected by leukapheresis prior to initiating standard concurrent RT and TMZ. Participants will receive the first and second infusions of EGFR BATs on days 14 and 21 after finishing concurrent RT and TMZ and then receive an infusion on day 21 of the first six cycles of TMZ.
  Interventions: Drug: EGFR BATs with TMZ following SOC RT/TMZ
- Subcohort for MGMT unmethylated patients (Experimental): Study participants will have cells collected by leukapheresis prior to initiating standard concurrent RT and TMZ. About 4 weeks after completion of RT/TMZ, participants will receive 8 weekly doses of EGFR BATs.
  Interventions: Drug: Weekly EGFR BATs following SOC RT/TMZ

INTERVENTIONS:
Drug: EGFR BATs with TMZ following SOC RT/TMZ — Standard of care: 6 weeks of RT and TMZ and 6 cycles of TMZ (150-200 mg/m2) on days 1-5 of each 28 day cycle Experimental: EGFR BATs 2 and 3 weeks after completing RT, and then on day 21 of each cycle of TMZ.
  Arms: Main Study
Drug: Weekly EGFR BATs following SOC RT/TMZ — Standard of care: 6 weeks of RT and TMZ Experimental: 8 weekly doses of EGFR BATs following SOC RT and TMZ
  Arms: Subcohort for MGMT unmethylated patients

SUMMARY:
This is a phase I trial using EGFR Bi-armed Activated T-cells (BATs) in combination with standard of care temozolomide (TMZ) and radiation (RT) in patients with glioblastoma (GBM). The purpose of the study is to determine a safe dose of EGFR BATs when given with standard of care therapy.

DETAILED DESCRIPTION:
In addition to finding the safe dose of EGFR BATs, immune evaluations will be performed as delineated in the schedule of events to measure immune responses during all stages of treatment for GBM.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically-confirmed newly diagnosed intracranial GBM or gliosarcoma
2. Age ≥ 18 years.
3. Karnofsky Performance Status ≥ 60.
4. Be willing and able to provide written informed consent for the trial.
5. For patients with resection, CT/MRI with contrast must be performed within 72 hours following resection. Intraoperative post resection MRI is acceptable. No post surgery CT/MRI is required for patients who have received biopsy.
6. Females of childbearing potential, and males, must be willing to use an effective method of contraception
7. Females of childbearing potential should have a negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
8. Demonstrate adequate organ function as defined below. All screening labs should be performed within 10 days prior to apheresis.

Absolute lymphocyte count ≥ 500/mm3, Absolute neutrophil count (ANC) ≥1,000 /mcL, Platelets ≥ 100,000 / mcL, Hemoglobin ≥ 9 g/dL (or ≥5.6 mmol/L without transfusion or EPO dependency (within 7 days of assessment), BUN ≤ 1.5 X upper limit of normal (ULN), Serum creatinine within the normal limits OR Measured or calculated creatinine clearance ≥60 mL/min/1.73m2, Serum total bilirubin ≤ 1.5 X ULN OR AST (SGOT) and ALT (SGPT) ≤ 5 X ULN, Albumin >2.5 mg/dL, International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X ULN, unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants

i. Additional inclusion criteria for sub-cohort: MGMT unmethylated according to UVA pathology testing

Exclusion Criteria:

1. Patients with a diagnosis of another malignancy within 3 years of being on-study. Exceptions include basal cell carcinoma of the skin, or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer. Patients must not be on any treatment for another malignancy.
2. Patients with evidence of leptomeningeal dissemination or subependymal spread on initial MRI.
3. Patients with extracranial metastases.
4. Known hypersensitivity to cetuximab or other EGFR antibody.
5. Alpha 1,3 Galactose IgE ("alpha gal") test result outside of the reference range (indicating likely hypersensitivity to cetuximab)
6. Evidence of active bleeding or bleeding diathesis.
7. Cardiac Status: Patients will be ineligible for treatment on this protocol if (prior to protocol entry):

   There is a history of a recent (within one year) myocardial infarction or stroke.

   There is a current or prior history of angina/coronary symptoms requiring medications and/or evidence of depressed left ventricular function (LVEF < 45% by MUGA or ECHO).

   There is clinical evidence of congestive heart failure requiring medical management (irrespective of MUGA or ECHO results).
8. Has Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies) or known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
9. Has received a live vaccine within 30 days of planned start of study therapy.
10. Has received any treatment for GBM besides surgery.
11. Females must not be breastfeeding.
12. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
13. A patient may be excluded if, in the opinion of the treating clinician, the patient is not capable of being compliant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-12-08 (Actual); Study Completion 2023-05-08 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | The study will not advance to the next dose until 7 days after the last patient in the cohort completes his or her second infusion of EGFR BATs
  Maximum tolerated dose will be based on number of dose limiting toxicities at each dose level

SECONDARY OUTCOMES:
Immune measures in blood- cellular phenotype | Before surgery (optional), during screening, at apheresis, at multiple timepoints during study treatment, following completion of study treatment, and every 2-6 months after completion of EGFR BATs infusions through 1 year after last EGFR BATs infusion
  Sequential monitoring of cellular phenotype
Immune measures in blood- interferon-γ | Before surgery (optional), during screening, at apheresis, at multiple timepoints during study treatment, following completion of study treatment, and every 2-6 months after completion of EGFR BATs infusions through 1 year after last EGFR BATs infusion
  Sequential monitoring of interferon-γ
Immune measures in blood- EliSpots | Before surgery (optional), during screening, at apheresis, at multiple timepoints during study treatment, following completion of study treatment, and every 2-6 months after completion of EGFR BATs infusions through 1 year after last EGFR BATs infusion
  Sequential monitoring of EliSpots
Immune measures in blood- anti-GBM cytotoxicity of peripheral blood mononuclear cells directed at GBM cell lines | Before surgery (optional), during screening, at apheresis, at multiple timepoints during study treatment, following completion of study treatment, and every 2-6 months after completion of EGFR BATs infusions through 1 year after last EGFR BATs infusion
  Sequential monitoring of anti-GBM cytotoxicity of peripheral blood mononuclear cells directed at GBM cell lines
Immune measures in blood- serum cytokine patterns | Before surgery (optional), during screening, at apheresis, at multiple timepoints during study treatment, following completion of study treatment, and every 2-6 months after completion of EGFR BATs infusions through 1 year after last EGFR BATs infusion
  Sequential monitoring of serum cytokine patterns
Immune measures in blood- anti-GBM antibodies | Before surgery (optional), during screening, at apheresis, at multiple timepoints during study treatment, following completion of study treatment, and every 2-6 months after completion of EGFR BATs infusions through 1 year after last EGFR BATs infusion
  Sequential monitoring of anti-GBM antibodies
Clinical response | Every 3 months following last study visit until death or study closure, expected within 5 years
  Progression-free survival (PFS)
Survival | Every 3 months following last study visit until death or study closure, expected within 5 years
  Overall Survival (OS)
Response Rate | Every 3 months following last study visit until death or study closure, expected within 5 years
  Objective Response Rate
Correlation of imaging to PFS and OS | Up to 12 months after study treatment completion
  Imaging (extent of resection) will be evaluated for correlation with PFS and OS.
Correlation of pathology to PFS and OS | Up to 12 months after study treatment completion
  EGFR expression and tumor-infiltrating lymphocytes and age will be evaluated for correlation with PFS and OS.
Correlation of clinical response to PFS and OS | Up to 12 months after study treatment completion
  Steroid use at the time of leukapheresis and age will be evaluated for correlation with PFS and OS.
Correlation of immune response to PFS and OS | Up to 12 months after study treatment completion
  Immune response characteristics will be evaluated for correlation with PFS and OS.
Adverse events, including dose limiting toxicities | Through 30 days following last dose of EGFR BATs
  Safety of 8 weekly doses of BATs in unmethylated MGMT patients without adjuvant temozolomide

CONTACTS AND LOCATIONS:
Overall Officials: Camilo Fadul, MD, Principal Investigator — University of Virginia
Locations (1):
- Samantha Brooks, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lum LG, Thakur A, Al-Kadhimi Z, Colvin GA, Cummings FJ, Legare RD, Dizon DS, Kouttab N, Maizel A, Colaiace W, Liu Q, Rathore R. Targeted T-cell Therapy in Stage IV Breast Cancer: A Phase I Clinical Trial. Clin Cancer Res. 2015 May 15;21(10):2305-14. doi: 10.1158/1078-0432.CCR-14-2280. Epub 2015 Feb 16. PMID 25688159
- [Background] Vaishampayan U, Thakur A, Rathore R, Kouttab N, Lum LG. Phase I Study of Anti-CD3 x Anti-Her2 Bispecific Antibody in Metastatic Castrate Resistant Prostate Cancer Patients. Prostate Cancer. 2015;2015:285193. doi: 10.1155/2015/285193. Epub 2015 Feb 23. PMID 25802762
- [Derived] Fadul CE, Thakur A, Kim J, Kassay-McAllister J, Schalk D, Lopes MB, Donahue J, Purow B, Dillon P, Le T, Schiff D, Liu Q, Lum LG. Phase I study targeting newly diagnosed grade 4 astrocytoma with bispecific antibody armed T cells (EGFR BATs) in combination with radiation and temozolomide. J Neurooncol. 2024 Jan;166(2):321-330. doi: 10.1007/s11060-024-04564-y. Epub 2024 Jan 23. PMID 38263486